CLINICAL TRIAL: NCT01447407
Title: Phase 1b Study to Evaluate the Safety and Immunogenicity of NDV-3 Formulated With or Without Alum (AlOH) and Administered Either Intramuscular (IM) or Intradermally (ID) to Healthy Adults
Brief Title: Effect of Adjuvant & Route of Administration on Safety & Immunogenicity of NDV-3 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NovaDigm Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NDV3-002
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Staphylococcal Infections; Yeast Infections; Candidiasis
Keywords: Staphylococcal infections; Yeast infections; Candidiasis
MeSH Terms: conditions — Staphylococcal Infections; Candidiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- NDV-3 vaccine with alum IM (Active Comparator): 300 ug Als3 and 0.5 mg Al as alum in PBS per dose, one dose administered IM
  Interventions: Biological: NDV-3 vaccine with alum IM
- NDV-3 vaccine without alum IM (Active Comparator): 300 ug Als3 in PBS per dose, one dose administered IM
  Interventions: Biological: NDV-3 vaccine without alum IM
- Placebo IM (Placebo Comparator): 0.5 mg Al as alum in PBS per dose, one dose administered IM
  Interventions: Biological: Placebo with alum IM
- NDV-3 vaccine without alum ID (Active Comparator): 30 ug Als3 in PBS per dose, one dose administered ID
  Interventions: Biological: NDV-3 vaccine without alum ID

INTERVENTIONS:
Biological: NDV-3 vaccine with alum IM — One dose administered IM
  Arms: NDV-3 vaccine with alum IM
Biological: NDV-3 vaccine without alum IM — One dose administered IM
  Arms: NDV-3 vaccine without alum IM
Biological: Placebo with alum IM — One dose administered ID
  Arms: Placebo IM
Biological: NDV-3 vaccine without alum ID — One dose administered ID
  Arms: NDV-3 vaccine without alum ID

SUMMARY:
This partially-blind, placebo controlled study is a Phase 1b study using an investigational vaccine, NDV-3, directed against Staphylococcus aureus and Candida sp. This study will compare NDV-3 administered with or without alum delivered intramuscularly (IM) at one dose level. It will also evaluate a lower dose of NDV-3 without alum delivered intradermally (ID) compared to placebo delivered ID.

DETAILED DESCRIPTION:
Preclinical studies in mice have established that several members of the Als family of proteins induce a protective immune response in mice and allow high survival rates following challenge with highly virulent doses of either Candida or S. aureus. Als3 (the antigen in the NDV-3 investigational vaccine) is the most effective member of the Als protein family in protecting mice from challenge with either Candida or S. aureus. The first Phase 1 study enrolled 40 healthy subjects that received placebo (N=10), 1 dose (N=30) or 2 doses (N=19) of the NDV-3 vaccine administered intramuscularly (IM). The vaccine was well tolerated and highly immunogenic. This study will evaluate the safety, tolerability and immunogenicity of one dose of NDV-3 vaccine formulated with and without alum given IM and also a lower dose without alum given intradermally (ID). Subjects will have follow-up visits to assess the safety tolerability and immune responses at selected time points up to 90 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent document prior to screening. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English.
2. Completed the screening process (as described in this protocol) within 28 days prior to dosing.
3. Healthy male and female volunteers 18-50 years of age, inclusive, at the time of dosing.
4. No clinically significant deviation from normal as judged by the investigator(s) in the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations.
5. Female volunteers must be one of the following:

   * of childbearing potential and practicing an acceptable method of birth control as judged by the Investigator(s)
   * naturally postmenopausal (no menses) for at least 1 year and has a documented FSH level ≥ 40 mIU/mL
   * surgically postmenopausal (bilateral oophorectomy or hysterectomy)
   * sterile (surgically [bilateral tubal ligation] or the Essure® Procedure) Female volunteers that are surgically sterile or surgically postmenopausal must provide documentation of the bilateral tubal ligation, bilateral oophorectomy, or hysterectomy prior to dosing or the volunteer must agree to use a medically acceptable method of birth control. The Essure® Procedure must have been inserted at least 3 months prior with documentation of the Essure® confirmation test prior to Period I dosing. If the procedure was inserted less than 3 months prior to Period I dosing or proper documentation of the confirmation test is not provided, the volunteer must agree to use an additional medically acceptable method of birth control.

Exclusion Criteria:

1. Reports receiving any investigational drug, investigational vaccine, or investigational device within 30 days prior to dosing.
2. Reports any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the Investigator(s).
3. Clinical laboratory test values outside the accepted range.
4. When confirmed upon additional testing, demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
5. Demonstrates a positive drug screen for non-prescription drugs.
6. Reports a clinically significant illness during the 28 days prior to dosing (as determined by the Investigator[s]).
7. Reports a history of allergic response(s) to nickel or anaphylaxis (or other serious reactions) to aluminum.
8. Reports receiving any live attenuated vaccine including FluMist® within 6 weeks prior to dosing or any licensed inactivated vaccine within 3 weeks prior to dosing.
9. Reports the use of any immunosuppressive drugs, including systemic corticosteroids, within 4 weeks prior to dosing.
10. Reports the use of any medications or treatments that may alter immune responses to the study vaccine within 3 weeks prior to dosing (eg, cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin [BCG], monoclonal antibodies, radiation therapy).
11. Reports a history of clinically significant allergies including food or drug allergies or anaphylaxis (or other serious reactions) to vaccines.
12. Reports a history of drug or alcohol addiction or abuse within the past year.
13. Reports receiving any blood products within 3 months prior to dosing and throughout the study.
14. Reports donating blood within 28 days prior to dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
15. Reports donating plasma (e.g. plasmapheresis) within 14 days prior to dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
16. Demonstrates, in the opinion of study staff, veins unsuitable for repeated venipuncture (e.g. veins difficult to locate, access, or puncture; veins with a tendency to rupture during or after puncture).
17. Pregnant, lactating, breastfeeding, or intends to become pregnant over the course of the study.
18. Demonstrates a positive pregnancy screen.
19. Reports smoking or using tobacco products or is currently using nicotine products (patches, gums, etc). Thirty (30) days abstinence prior to dosing is required.
20. Any other medical and/or social (e.g. uncooperative or non-compliant) reason which, in the opinion of the investigator(s), would prevent participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research Clinical Site, Fargo, North Dakota, United States

REFERENCES:
- [Background] Schmidt CS, White CJ, Ibrahim AS, Filler SG, Fu Y, Yeaman MR, Edwards JE Jr, Hennessey JP Jr. NDV-3, a recombinant alum-adjuvanted vaccine for Candida and Staphylococcus aureus, is safe and immunogenic in healthy adults. Vaccine. 2012 Dec 14;30(52):7594-600. doi: 10.1016/j.vaccine.2012.10.038. Epub 2012 Oct 22. PMID 23099329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects withdrew before completing Day 28 and were replaced. One subject withdrew before the last visit. While this subject is not considered to have completed the study, data from this subject are included in the immunogenicity and culture results.
Groups:
- NDV-3 Vaccine With Alum: NDV-3 (300 ug Als3) vaccine with alum administered IM: One dose administered IM
- NDV-3 Vaccine Without Alum: NDV-3 (300 ug Als3) vaccine without alum administered IM: One dose administered IM
- Placebo: Placebo administered ID: One dose saline placebo administered ID
- NDV-3 Vaccine ID: NDV-3 (30 ug Als3) vaccine without alum administered ID: One dose administered ID
Period: Overall Study
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Started | 41 | 40 | 41 | 42
Completed | 39 | 40 | 40 | 40
Not Completed | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID | Total
Number analyzed (Participants) | 41 | 40 | 41 | 42 | 164
Age, Continuous [Mean (Full Range); unit: years] | 31.8 [18 to 47] | 30.1 [18 to 49] | 32.3 [19 to 50] | 31.0 [18 to 50] | 31.3 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 34 | 34 | 134
  Male | 8 | 7 | 7 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 41 | 40 | 41 | 41 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 4
  White | 38 | 37 | 36 | 38 | 149
  More than one race | 3 | 1 | 3 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The primary objective of this study is to assess the safety of a single dose of NDV-3 vaccine, administered either IM with or without alum adjuvant at one dose level or ID at a lower dose level, compared to placebo. Clinical evaluations will be assessed on each subject at selected time points up to 90 days post-vaccination.
Time Frame: Up to 90 days post-vaccination
Population: All subjects completing study. Additionally, a subject in Group 4 withdrew from the study before the very last visit, so while this subject is not considered to have completed the study, immunogenicity and culture data for this subject were included.
Measure: Number; unit: participants
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
participants
  >=1 TEAE | 35 | 33 | 30 | 36
  >=1 severe TEAE | 2 | 0 | 4 | 2
  >=1 severe drug-related TEAE | 0 | 0 | 0 | 0
  DIscontinued for >=1 TEAE | 0 | 0 | 0 | 0

2. Secondary Outcome: Immunogenicity - Serum Anti-Als3 IgG
Description: A secondary objective is to compare the serum IgG immune response between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. Serum IgG will be evaluated by ELISA on serial-diluted samples, resulting in titer values of reciprocal dilution at which the ELISA readout is three times greater than the assay background value.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Titer
  Baseline | 372 (3.12) | 320 (3.07) | 363 (2.93) | 375 (3.53)
  Day 7 | 4447 (6.31) | 3070 (6.71) | 365 (2.81) | 874 (5.25)
  Day 14 | 44675 (3.04) | 22675 (6.58) | 370 (2.89) | 5153 (6.97)
  Day 28 | 38898 (2.83) | 19220 (6.00) | 377 (2.93) | 4513 (6.60)
  Day 90/Exit | 20853 (3.24) | 11771 (5.93) | 347 (2.71) | 3282 (5.55)

3. Secondary Outcome: Immunogenicity - Serum Anti-Als3 IgA1
Description: A secondary objective is to compare the serum IgA1 immune response between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. Serum IgA1 will be evaluated by ELISA on serial-diluted samples, resulting in titer values of reciprocal dilution at which the ELISA readout is three times greater than the assay background value.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Titer
  Baseline | 573 (4.07) | 480 (3.44) | 418 (3.72) | 550 (4.93)
  Day 7 | 7643 (6.61) | 5497 (7.01) | 431 (3.69) | 1640 (6.56)
  Day 14 | 69616 (3.1) | 34946 (6.77) | 429 (3.93) | 9356 (6014)
  Day 28 | 43790 (2.59) | 19999 (5.36) | 412 (3.86) | 7400 (6.33)
  Day 90/Exit | 20656 (2.51) | 10698 (4.61) | 404 (3.78) | 3641 (5.18)

4. Secondary Outcome: Immunogenicity - Cervicovaginal Wash Anti-Als3 IgG
Description: A secondary objective is to compare the cervicovaginal wash IgG immune response between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. Cervicovaginal wash IgG will be evaluated by ELISA on serial-diluted samples, resulting in titer values of reciprocal dilution at which the ELISA readout is three times greater than the assay background value.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Titer
  Baseline | 2 (1.5) | 2 (1.55) | 3 (2.12) | 3 (1.98)
  Day 7 | 4 (3.98) | 6 (5.84) | 2 (1.61) | 3 (2.45)
  Day 14 | 78 (7.12) | 26 (7.50) | 3 (1.99) | 8 (4.27)
  Day 28 | 44 (5.85) | 26 (7.09) | 3 (2.20) | 8 (4.63)
  Day 90/Exit | 20 (4.93) | 13 (4.65) | 3 (2.11) | 6 (4.35)

5. Secondary Outcome: Immunogenicity - Cervicovaginal Wash Anti-Als3 IgA1
Description: A secondary objective is to compare the cervicovaginal wash IgA1 immune response between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. Cervicovaginal wash IgA1 will be evaluated by ELISA on serial-diluted samples, resulting in titer values of reciprocal dilution at which the ELISA readout is three times greater than the assay background value.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Titer
  Baseline | 3 (2.03) | 3 (2.08) | 3 (2.24) | 3 (2.5)
  Day 7 | 5 (2.87) | 7 (6.64) | 3 (1.45) | 4 (2.71)
  Day 14 | 83 (4.50) | 29 (6.48) | 3 (1.64) | 12 (4.23)
  Day 28 | 36 (3.82) | 25 (6.72) | 3 (2.40) | 8 (4.56)
  Day 90/Exit | 15 (3.18) | 8 (3.27) | 3 (1.98) | 5 (3.40)

6. Secondary Outcome: Immunogenicity - Number of Participants Positive for Peripheral Blood Mononuclear Cells (PBMCs) Producing Als3-specific Interferon-gamma (IFN-g)
Description: A secondary objective is to compare the cellular immune response for Als3-specific production of IFN-g from PBMCs between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. The IFN-g cellular immune responses will be evaluated by ELISpot using approximately 200,000 PBMCs per well. A positive response was defined as a sample with greater than 20 spot forming units per 10^6 PBMCs.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Count of Participants; unit: Participants
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Participants
  Baseline | 7 | 9 | 7 | 5
  Day 7 | 27 | 25 | 10 | 20
  Day 14 | 19 | 21 | 5 | 20
  Day 90/Exit | 25 | 18 | 9 | 14

7. Secondary Outcome: Immunogenicity - Number of Participants Positive for Peripheral Blood Mononuclear Cells (PBMCs) Producing Als3-specific Interleukin-17A (IL-17A)
Description: A secondary objective is to compare the cellular immune response for Als3-specific production of IL-17A from PBMCs between the 2 dose levels, routes of administration, and effects of alum adjuvant, at selected time points up to 90 days post-vaccination. The IL-17A cellular immune responses will be evaluated by ELISpot using approximately 200,000 PBMCs per well. A positive response was defined as a sample with greater than 20 spot forming units per 10^6 PBMCs.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 90/Exit
Measure: Count of Participants; unit: Participants
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
Number analyzed (Participants) | 39 | 40 | 40 | 40
Participants
  Baseline | 6 | 10 | 12 | 9
  Day 7 | 22 | 19 | 8 | 13
  Day 14 | 15 | 17 | 7 | 16
  Day 90/Exit | 17 | 15 | 18 | 23

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | NDV-3 Vaccine With Alum | NDV-3 Vaccine Without Alum | Placebo | NDV-3 Vaccine ID
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 35/41 | 33/40 | 30/41 | 36/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NDV-3 Vaccine With Alum (N=41) | NDV-3 Vaccine Without Alum (N=40) | Placebo (N=41) | NDV-3 Vaccine ID (N=42)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 7 (7)
Fatigue (General disorders) | 4 (4) | 4 (4) | 4 (4) | 13 (13)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (8)
Injection site pain (General disorders) | 32 (32) | 18 (18) | 3 (3) | 15 (15)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (8)
Injection site swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 1 (1) | 5 (5) | 6 (6)
Protein total decreased (Investigations) | 2 (2) | 8 (8) | 3 (3) | 7 (7)
Protein urine present (Investigations) | 4 (4) | 0 (0) | 4 (4) | 4 (4)
Red blood cells urine positive (Investigations) | 5 (5) | 7 (7) | 9 (9) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 8 (8)
Headache (Nervous system disorders) | 10 (10) | 7 (7) | 9 (9) | 19 (19)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes